CLINICAL TRIAL: NCT03345277
Title: Continuous Temperature Measurement for Syndromic Surveillance
Status: Withdrawn | Type: Observational
Why Stopped: Study never reached the enrolling phase and PI has since relocated
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: AMK-2016.065
Record Dates: First submitted 2017-11-05; First posted 2017-11-17 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Continuous Temperature; Syndromic Surveillance; Long-term Care
Keywords: Termperature; Fever; Vital Signs
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous Temperature monitoring: All residents of a long-term care facility will be considered for the study over the predetermined timeframe. Residents who choose not to participate or are determined, by their care providers, to be inappropriate for inclusion will be excluded.
  Interventions: Other: Continuous Temperature monitoring

INTERVENTIONS:
Other: Continuous Temperature monitoring — Residents in a long term care facility will wear a thermometer continuously for 3 months, measuring their body temperature

SUMMARY:
Is it possible to detect infection before it is clinically apparent? Fever is one indicator of infection. However, until recently, continuous temperature monitoring has not been feasible. With the advent of microelectronics, long battery life, and wireless transmission, it is now possible to continuously measure, record and report body temperature. For a period of 90 days, residents of a long-term care facility will have their body temperature monitored and then those measurements will then be compared against other available healthcare data such as other recorded vital signs, nursing notes, provider visits, antibiotics, and hospitalization records for correlation of underlying infection.

DETAILED DESCRIPTION:
Over 1.5 million people live in 16,000 nursing homes (NH) in the USA and experience an average of 2 million infections a year. It is well known that NH residents are at risk of infection because of frequent hospital stays, advanced age, exposure to multiple courses of antibiotics, numerous comorbidities, diminished immune response, malnutrition, and cognitive impairment. The most common are pneumonia, UTIs, diarrheal illnesses, and skin and soft tissue infections. Infections in NH residents have been associated with adverse clinical outcomes, including high rates of morbidity and mortality, re-hospitalization, prolonged hospital stays and substantial healthcare expenses.

The identification of fever is a key component in the detection of infections. Studies have shown that standard definition for fever, 100.5 degrees F, is not sensitive to identify infections in elderly populations. The recommendation therefore is a fever of 99 degrees F or an increase of 2.4 degrees F from baseline. These changes in temperatures are also a significant indication that infection is present.

The collection of episodic temperatures in nursing home residents is challenging. The collection of baseline measurements for all residents is logistically unachievable. The continuous measurement of body temperature in any mobile population would be nearly impossible by any clinically standard means.

With the advent of microelectronics, long battery life, and wireless transmission, it is now possible to continuously measure, record and report body temperature.

What remains unknown is the feasibility and clinical utility of obtaining these measurements.

Therefore it is proposed that for a period of three months, residents of a single, long-term care facility have a wearable, thermometer applied to their skin. The medical-grade adhesive and thermometer will be changed every 2-3 days. The thermometer will provide continuous temperature measurement that will be sent wirelessly via Bluetooth to access points positioned throughout the facility.

The temperatures are reported wirelessly every minute and stored in a secure server. All participants and care providers are blinded to the temperature readings.

At the conclusion of the monitoring period, the temperature readings will be compared to the longitudinal healthcare record for each of the participants. Particular attention will be toward hospitalizations, antibiotics, nursing records, and clinic visits to determine episodes of infectious illness.

ELIGIBILITY:
Inclusion Criteria:

* Residents of a long-term care facility

Exclusion Criteria:

* Residents who choose not to participate or are determined, by their care providers, to be inappropriate for inclusion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents in a long term care facility.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Continuous temperature monitoring | 90 days duration for study participation
  monitoring temperature wirelessly via Bluetooth thermometer

CONTACTS AND LOCATIONS:
Overall Officials: Vernon Smith, MD, Principal Investigator — Avera Health
Locations (1):
- Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota, United States